CLINICAL TRIAL: NCT02263547
Title: Rapid Elimination Procedure of Teriflunomide With Colestipol Hydrochloride
Acronym: TERCOL
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: PK time points were not being met as expected. Determination that risks outweighed benefit.
Sponsor: Derrick Scott Robertson (Other)
Collaborators: Genzyme, a Sanofi Company (Industry); University of South Florida (Other)
Responsible Party: Sponsor-Investigator, Derrick Scott Robertson, Assistant Professor, University of South Florida
Organization: University of South Florida (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: GZ-2013-11023
Record Dates: First submitted 2014-09-30; First posted 2014-10-13 (Estimated); Results first posted 2019-07-01 (Actual); Last update posted 2020-04-03 (Actual); Status verified 2020-04

CONDITIONS: Teriflunomide Elimination; Healthy Volunteers
Keywords: teriflunomide; colestipol hcl
MeSH Terms: interventions — teriflunomide; Colestipol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- teriflunomide elimination with colestipol (Other)
  Interventions: Drug: teriflunomide; Drug: Colestipol

INTERVENTIONS:
Drug: teriflunomide
  Other Names: Aubagio
Drug: Colestipol

SUMMARY:
Primary Objective To determine if colestipol hydrochloride tablets can accelerate the elimination of teriflunomide. Teriflunomide will be administered for 14 days followed by colestipol dosing of 11 days. Total duration of the study is 40 days.

Secondary Objectives To collect information on the pattern of side effects with use of colestipol hydrochloride after teriflunomide administration and to determine the best duration of therapy needed for adequate elimination

DETAILED DESCRIPTION:
participants will be followed for 40 days to allow for time to administer a loading dose of teriflunomide and observe the elimination of that drug using colestipol hcl.

ELIGIBILITY:
Inclusion Criteria:

To be eligible for entry into this study, candidates must meet all of the following eligibility criteria at the time of the baseline visit:

1. Participants having provided informed consent with signature on informed consent form: the informed consent process should be complete with full discussion of all requirements and possible risks.
2. Healthy volunteer*
3. Aged 18-45 years, inclusive
4. Body Mass Index of 18-29 kg/m2 (body weight of 40-85 kg for women and 50-95 kg for men) *Healthy volunteer is defined as free of concomitant medications and use of either treatment, as deemed by the Investigator, is not contraindicated with any past medical history of the participant.

Exclusion Criteria:

1. Current smoker or past history as smoker.
2. Unable to provide informed consent to participate in the study Such as a mental condition rendering the participant unable to understand the nature, scope, and possible consequences of the study
3. Participant unlikely to comply with protocol as determined by Investigator, eg, uncooperative attitude, inability to return for follow-up visits
4. Clinically relevant cardiovascular, hepatic, neurological, endocrine, or other major systemic disease making implementation of the protocol or interpretation of the study results difficult or that would put the participant at risk by participating in the study
5. Persistent significant or severe infection, either acute or chronic
6. Recent history of drug or alcohol abuse within that past 6 months (participants will be asked to refrain from alcohol and drug use during the course of the study)
7. Participant is the Investigator or any Sub-investigator, research assistant, pharmacist, study coordinator, other staff or relative thereof, directly involved in the conduct of the protocol
8. Prior use of any investigational drug in the preceding 6 months
9. Liver function impairment or persisting elevations (confirmed by retest) of alanine aminotransferase (ALT), aspartate aminotransferase (AST), or direct bilirubin greater than 2x the upper limit of normal range (ULN).
10. Pregnant or breast-feeding women or those who plan to become pregnant during the study
11. Women of childbearing potential not protected by effective contraceptive method of birth control and/or who are unwilling or unable to be tested for pregnancy.
12. Participants wishing to parent children (be a partner in the conception of a child) during the course of the trial.
13. Participants with significantly impaired bone marrow function or significant anemia, leukopenia, or thrombocytopenia (confirmed by retest):

    * Hematocrit < 35% and/or
    * Absolute white blood cell count < 3000 cells/mm3 (μL) and/or
    * Platelet count < 150 000 cells/mm3 (μL) and/or- Absolute neutrophil ≤ 1500 cells/mm3 (μL)
14. Any known history of severe preexisting constipation
15. History of swallowing disorder or difficulty swallowing

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 14 (Actual)
Dates: Start 2015-03; Primary Completion 2016-06 (Actual); Study Completion 2016-06 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- USF Carol and Frank Morsani Center for Advanced Healthcare, Tampa, Florida, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Enrollment occurred from March 2015 through May 2016 at the USF Carol and Frank Morsani Center.
Pre-assignment Details: Participants were healthy individuals with no significant health history or concomitant medication use.
Groups:
- Teriflunomide Elimination With Colestipol: teriflunomide
  Colestipol
Period: Overall Study
Arm/Group | Teriflunomide Elimination With Colestipol
Started | 14
Completed | 11
Not Completed | 3
Not completed — Adverse Event | 1
Not completed — Lost to Follow-up | 2

BASELINE CHARACTERISTICS:
Arm/Group | Teriflunomide Elimination With Colestipol
Number analyzed (Participants) | 14
Age, Continuous [Mean (Standard Deviation); unit: years] | 24.5 (7.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 10
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Caucasian | 7
  Black | 2
  Asian | 1
  Hispanic | 4
BMI [Mean (Standard Deviation); unit: kg/m^2] | 23.9 (2.7)

OUTCOME MEASURES:

1. Primary Outcome: Primary Outcome Measures: Teriflunomide Concentrations at Day 28
Description: After receiving 14 days of teriflunomide, participants will take 11 days of colestipol to wash out the teriflunomide (measuring the levels of teriflunomide in the blood at each visit)
Time Frame: 28 days after the start in the study
Measure: Mean (Standard Deviation); unit: teriflunomide level (mcg/ml)
Arm/Group | Teriflunomide Elimination With Colestipol
Number analyzed (Participants) | 14
teriflunomide level (mcg/ml) | 9.36 (4.26)

2. Secondary Outcome: Secondary Outcome Measure: Mean Percentage Change of Serum Teriflunomide Levels Percentage Change of Teriflunomide Concentrations at Day 8, Day 14, Day 26 ad Day 36 Following Administration of Colestipol Hydrochloride Tablets.
Description: The last blood draw will be about 50 days from the start of the study
Time Frame: duration of study about 50 days
Measure: Mean (Standard Deviation); unit: percentage change in teriflunomide level
Arm/Group | Teriflunomide Elimination With Colestipol
Number analyzed (Participants) | 14
percentage change in teriflunomide level
  8 days after colestipol hcl administered | -56.4 (21.9)
  14 days after colestipol hcl administered | -74.9 (27)
  26 days after colestipol hcl administered | -94.9 (6.3)
  36 days after colestipol hcl administered | -96.9 (3.7)

ADVERSE EVENTS:
Arm/Group | Teriflunomide Elimination With Colestipol
Serious Adverse Events (participants affected / at risk) | 0/14
Other Adverse Events (participants affected / at risk) | 12/14
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Teriflunomide Elimination With Colestipol (N=14)
Anticipated Adverse events (Gastrointestinal disorders) | 11 (11) — nausea, diarrhea, abdominal discomfort, heartburn
Upper Respiratory Infection (Infections and infestations) | 4 (4)

LIMITATIONS AND CAVEATS:
small number of subjects analyzed with some lost to followup

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less